CLINICAL TRIAL: NCT04904458
Title: The Effects of the "Enfacement Illusion" on Pain Perception in Patients Suffering From Chronic Migraine.
Brief Title: Enfacement Illusion and Chronic Migraine Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Enfacement Illusion2020
Record Dates: First submitted 2021-05-05; First posted 2021-05-27 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-05

CONDITIONS: Migraine
Keywords: Virtual reality; Chronic migraine; Pain; Enfacement illusion; Non-pharmacological treatments; Emotional regulation
MeSH Terms: conditions — Migraine Disorders; Pain; Emotional Regulation | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group receives the Enfacement Illusion toward a happy emotional face through a head mounted display.
  Interventions: Other: Experimental group ("enfacement illusion")
- Control Group (Sham Comparator): The control group receives the exposure to a pleasant virtual environment through a head mounted display
  Interventions: Other: Control Group (Pleasant virtual environment exposure)

INTERVENTIONS:
Other: Experimental group ("enfacement illusion") — Virtual reality enfacement illusion exposure
  Arms: Experimental group
Other: Control Group (Pleasant virtual environment exposure) — Pleasant virtual environment exposure
  Arms: Control Group

SUMMARY:
The concept of body image can be described as "the intentional content of consciousness comprising perceptions, attitudes and beliefs relating to one's body". Over the years, there has been a growing interest in this topic, highlighting that body image can be distorted in people suffering from pain conditions, especially in the case of chronic pain. One way of modulating the perception of pain through the perception of body image is through the use of interventions based on visual feedback. In this regard, some studies have highlighted the possibility of reducing the perception of pain in healthy and clinical populations with the use of "illusions" of one's own body created through immersive virtual reality. For example, through the use of synchronous visual-tactile multisensory stimulation on one's own face / body and on that of others (fake body), is possible to induce illusions of self-recognition in other fake bodies. In the case of the face, this type of illusion of belonging of other faces is commonly known as the "enfacement illusion", through which is possible to change or modulate the self-representation, with important implications for all those subjects who have distorted body representations, such as patients suffering from chronic pain. The main goal of the present protocol is to evaluate the effects of an experimental treatment based on enfacement illusion on the perception of pain (VAS scale) with respect to a control condition (pleasant virtual environment exposure). The secondary objective is to study any correlations between pain and body image, personal, clinical and psychological intrapersonal variables. One-hundred patients with chronic headache will be randomly assigned to the two conditions: experimental group (based on the "enfacement illusion") and control group (exposed to a pleasant virtual environment). Both conditions include an immersive virtual reality treatment of 3 sessions of 15 minutes each, during one week.

DETAILED DESCRIPTION:
The concept of body image can be described as "the intentional content of consciousness comprising perceptions, attitudes and beliefs relating to one's body". Over the years, there has been a growing interest in this topic, highlighting that body image can be distorted in people with pain, especially in the case of chronic pain. In the context of migraine, some studies have shown that the perception of pain can alter both the facial recognition capacity and the visuospatial perception compared to healthy subjects. Furthermore, other studies have shown that by reducing the altered perception of body image in patients with migraine associated with overuse of drugs, it is possible to induce beneficial effects on their affective state and on the perception of pain. One way to modify the perception of pain through the perception of the body image consists in the use of interventions based on visual feedback. Other studies have also highlighted the possibility of reducing the perception of pain in healthy and clinical populations with the use of "illusions" of one's body created through immersive virtual reality. In a pilot study conducted at IRCCS Mondino, the effect of different visual feedback conditions (facial expressions): positive, neutral, negative and white screen (control condition) on the modulation of pain perception in a sample of 38 patients with chronic migraine, demonstrated that the observation of a positive emotional face stimuli, when compared to other conditions, decreased their pain perception. Further, other studies demonstrated that the use of synchronous visual-tactile multisensory stimulation on one's face / body and on that of others (fake body) is able to induce illusions of self-recognition toward the others body part. This illusion of belonging of other faces thus created is known as "enfacement illusion" and seems to be positively correlated to the empathic traits of the subjects mediated by emotion regulation. Other studies show that the "enfacement illusion" seems to be a good strategy for changing the self-representation, with important implications for all those subjects who have distorted body representations, such as patients suffering from chronic pain. This study aims to evaluate whether through the "enfacement illusion" of representing oneself in a happy face exposed through an immersive virtual reality system (experimental group) it is possible to reduce the perception of pain in patients with chronic migraine. This effect would be mediated by an improved body image and empathy for positive emotions. In order to demonstrate the effects of the "enfacement illusion" on their own body representation and pain perception, a control group will be subjected to a positive exposure (pleasant environment) in an immersive virtual environment, which seems to be able to produce distracting effects on pain perception in patients with chronic migraine. It is hypothesized that patients with chronic migraine exposed to the "enfacement illusion" will experience greater pain relief and improve the perception of their body image compared to the control group. Therefore, the present study aims to show a possible relationship between the distortion of the body image and pain perception and, therefore, to demonstrate the effectiveness of the use of "enfacement illusion" as a cognitive behavioral intervention aimed at alleviating pain in clinical populations. Patients in the experimental group will be exposed to the "enfacement illusion" condition, conducted similarly to other studies. In detail, patients will see, through a virtual reality helmet, a virtual body sitting in front of them with a happy face expression. Each session will consist of three phases: (1) habituation to the virtual environment, (2) observation of the virtual facial expression, (3) multisensory stimulations (visuo-tactile stimulation).

Phase (1) habituation to the virtual environment: For approximately 2 minutes the experimenter will ask patients to describe what they see in the virtual environment, as well as the virtual body positioned in front of them.

Phase (2) observation of facial expression: the experimenter will ask patients to focus attention on the face of the virtual body sitting in front of them for about 1 minute.

Phase (3) multisensory with a brush. The multisensory (visual-tactile) stimulation is necessary to induce the sensation of belonging to the virtual body, and specifically to induce the sense of ownership toward the virtual face. The multisensory stimulation will last for 5 minutes.

The control group of this study, will be exposed to a visual stimulation by observing a pleasant immersive virtual reality environment for the duration of 5 minutes. As in the experimental group, in the first 2 minutes of immersion in the virtual environment, the experimenter will ask the patient to describe the virtual environment. Then, the patients will be immersed in the virtual environment for about 5 minutes.

In this frame, the primary goal of this double-blind randomized controlled trial is to assess whether the "enfacement illusion" of representing oneself (inducing the sense of ownership) in a happy face through an immersive virtual reality may reduce the perception of pain in patients with chronic migraine. A secondary goal is to evaluate the effects on the perception of one's body image and on the affective and emotional state of a treatment based on "enfacement illusion" with respect to a control condition. Both treatment protocols consist of 3 session/week, 15 minutes/day, of the virtual reality enfacement illusion exposure vs pleasant virtual environment exposure. Female patients with chronic migraine accomplishing the clinical characteristics included in the ICHD-III version for chronic migraine, with pain perception between 20 and 80 on a 0-100 visual analogue scale will be recruited from Headache Science center Unit of IRCCS Mondino Foundation.

All patients will undergo the following assessment measures:

Pre / post treatment (T0-T1): all subjects will be assessed as regards their affective and emotional state with: Body Satisfaction Scale (BSS), Hospital Anxiety and Depression Scale (HADS), Emotive Regulation Questionnaire (ERQ) , and the Difficulties in Emotion Regulation Scale (DERS), Pain-Visual Analogue Scale (VAS), Body Image Questionnaire (BIQ), and Positive and Negative Affect Schedule (PANAS).

Pre / post visual exposure session: all subjects will be assessed with the Pain-Visual Analogue Scale (VAS), Body Image Questionnaire (BIQ) and Positive and Negative Affect Schedule (PANAS).

After each visual exposure session: the patients of the experimental group will fill in a questionnaire relating to the level of sense of belonging (embodiment) of the virtual body. The control group will fill out a questionnaire relating to the level of immersion in the virtual environment.

ELIGIBILITY:
Inclusion Criteria:

1. Accomplish the clinical characteristics included in the ICHD-III version for chronic migraine.
2. Age between >18 to 65 year old (only women).
3. Previous history of migraine as primary headache.
4. Pain perception between 20 and 80 on a 0-100 VAS.

Exclusion Criteria:

1. Dementia, epilepsy, psychosis, mental retardation, pregnant and breastfeeding women.
2. Visual problems

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — There are studies reporting differences in pain perception between man and women (Wiesenfeld-Hallin, 2005)
Enrollment: 100 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Change fromT0 (baseline) toT1 (at the end of the intervention, i.e. after one-week)
  To assess the effects on pain perception measured by a 0-100 Visual Analogue Scale (VAS) of a one-week treatment based on "enfacement illusion" compared to a control condition (pleasant virtual environment exposure) in patients with chronic migraine

SECONDARY OUTCOMES:
Body Image Questionnaire (BIQ) | Change fromT0 (baseline) toT1 (at the end of the intervention, i.e. after one-week)
  To assess the effects on the perception of one's own body image and on the affective and emotional state of a one-week treatment based on "enfacement illusion" with respect to a control condition (pleasant virtual environment exposure). Pre / post each session all subjects will be evaluated with Body Image Questionnaire (BIQ). BIQ is a 19 -item questionnaire
Positive and Negative Affect Schedule (PANAS) | Change fromT0 (baseline) toT1 (at the end of the intervention, i.e. after one-week)
  To assess the effects on the perception of one's own body image and on the affective and emotional state of a treatment based on "enfacement illusion" with respect to a control condition (pleasant virtual environment exposure). Pre / post each session all subjects will be evaluated with Positive and Negative Affect Schedule (PANAS).
  Positive Affect Score: scores can range from 10 - 50, with higher scores representing higher levels of positive affect.
  Negative Affect Score: scores can range from 10 - 50, with lower scores representing lower levels of negative affect.
Body Satisfaction Scale (BSS) | Change fromT0 (baseline) toT1 (at the end of the intervention, i.e. after one-week)
  To assess the relationship between the affective and emotional state of patients and the change in the perception of pain and one's body image. Before and after the one-week treatment, all subjects will be assessed for what concerns their affective and emotional state with Body Satisfaction Scale (BSS).
The Hospital Anxiety and Depression Scale (HADS) | Change fromT0 (baseline) toT1 (at the end of the intervention, i.e. after one-week)
  To assess the relationship between the affective and emotional state of patients and the change in the perception of pain and one's body image. Before and after the one-week treatment, all subjects will be assessed for what concerns their affective and emotional state with the Hospital Anxiety and Depression Scale (HADS). The HADS questionnaire has seven items each for depression and anxiety subscales. Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression.
The Emotive Regulation Questionnaire (ERQ) | Change fromT0 (baseline) toT1 (at the end of the intervention, i.e. after one-week)
  To assess the relationship between the affective and emotional state of patients and the change in the perception of pain and one's body image. Before and after the one-week treatment, all subjects will be assessed for what concerns their affective and emotional state with the Emotive Regulation Questionnaire (ERQ). The Emotion Regulation Questionnaire (ERQ) is a 10-item self-report scale designed to assess habitual use of two commonly used strategies to alter emotion: cognitive reappraisal and expressive suppression.
The Difficulties in Emotion Regulation Scale (DERS) | Change fromT0 (baseline) toT1 (at the end of the intervention, i.e. after one-week)
  To assess the relationship between the affective and emotional state of patients and the change in the perception of pain and one's body image. Before and after the one-week treatment, all subjects will be assessed for what concerns their affective and emotional state with the Difficulties in Emotion Regulation Scale (DERS). The DERS is a 36-item self-report measure of six facets of emotion regulation. Items are rated on a scale of 1 ("almost never [0-10%]") to 5 ("almost always [91-100%]"). Higher scores indicate more difficulty in emotion regulation.
To assess the virtual reality experience within each treatment condition | Up to one-week
  After each treatment session, the patients of the experimental group will fill in a questionnaire relating to the level of sense of belonging (embodiment) of the virtual body. The control group will fill out a questionnaire relating to the level of immersion and presence in the virtual environment

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Tassorelli, Prof, Principal Investigator — Headache Science Center
Locations (1):
- Headache Science Center, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balzarotti, Stefania, Oliver P. John, and James J. Gross. 2010. "An Italian Adaptation of the Emotion Regulation Questionnaire." European Journal of Psychological Assessment. https://doi.org/10.1027/1015-5759/a000009.
- [Background] Costantini M, Musso M, Viterbori P, Bonci F, Del Mastro L, Garrone O, Venturini M, Morasso G. Detecting psychological distress in cancer patients: validity of the Italian version of the Hospital Anxiety and Depression Scale. Support Care Cancer. 1999 May;7(3):121-7. doi: 10.1007/s005200050241. PMID 10335929
- [Background] Longo MR, Schuur F, Kammers MP, Tsakiris M, Haggard P. What is embodiment? A psychometric approach. Cognition. 2008 Jun;107(3):978-98. doi: 10.1016/j.cognition.2007.12.004. Epub 2008 Feb 11. PMID 18262508
- [Background] Lotze M, Moseley GL. Role of distorted body image in pain. Curr Rheumatol Rep. 2007 Dec;9(6):488-96. doi: 10.1007/s11926-007-0079-x. PMID 18177603
- [Background] Matamala-Gomez M, Donegan T, Bottiroli S, Sandrini G, Sanchez-Vives MV, Tassorelli C. Immersive Virtual Reality and Virtual Embodiment for Pain Relief. Front Hum Neurosci. 2019 Aug 21;13:279. doi: 10.3389/fnhum.2019.00279. eCollection 2019. PMID 31551731
- [Background] Nicolodi M, Sandoval V. P012. Body image role in medication-overuse headache associated with persistent depressive disorder. J Headache Pain. 2015 Dec;16(Suppl 1):A111. doi: 10.1186/1129-2377-16-S1-A111. No abstract available. PMID 28132277
- [Background] Porciello G, Bufalari I, Minio-Paluello I, Di Pace E, Aglioti SM. The 'Enfacement' illusion: A window on the plasticity of the self. Cortex. 2018 Jul;104:261-275. doi: 10.1016/j.cortex.2018.01.007. Epub 2018 Feb 9. PMID 29478669
- [Background] Price DD, McGrath PA, Rafii A, Buckingham B. The validation of visual analogue scales as ratio scale measures for chronic and experimental pain. Pain. 1983 Sep;17(1):45-56. doi: 10.1016/0304-3959(83)90126-4. PMID 6226917
- [Background] Sforza A, Bufalari I, Haggard P, Aglioti SM. My face in yours: Visuo-tactile facial stimulation influences sense of identity. Soc Neurosci. 2010;5(2):148-62. doi: 10.1080/17470910903205503. Epub 2009 Oct 7. PMID 19813138
- [Background] Terracciano A, McCrae RR, Costa PT Jr. Factorial and construct validity of the Italian Positive and Negative Affect Schedule (PANAS). Eur J Psychol Assess. 2003;19(2):131-141. doi: 10.1027//1015-5759.19.2.131. PMID 20467578
- [Background] de Tommaso M, Calabrese R, Vecchio E, De Vito Francesco V, Lancioni G, Livrea P. Effects of affective pictures on pain sensitivity and cortical responses induced by laser stimuli in healthy subjects and migraine patients. Int J Psychophysiol. 2009 Nov;74(2):139-48. doi: 10.1016/j.ijpsycho.2009.08.004. Epub 2009 Aug 25. PMID 19712710
- [Background] Valentini E, Martini M, Lee M, Aglioti SM, Iannetti G. Seeing facial expressions enhances placebo analgesia. Pain. 2014 Apr;155(4):666-673. doi: 10.1016/j.pain.2013.11.021. Epub 2013 Dec 6. PMID 24315986
- [Background] Yetkin-Ozden S, Ekizoglu E, Baykan B. Face recognition in patients with migraine. Pain Pract. 2015 Apr;15(4):319-22. doi: 10.1111/papr.12191. Epub 2014 Apr 12. PMID 24725507
- [Background] Wiesenfeld-Hallin Z. Sex differences in pain perception. Gend Med. 2005 Sep;2(3):137-45. doi: 10.1016/s1550-8579(05)80042-7. PMID 16290886